CLINICAL TRIAL: NCT06877468
Title: Developing Tailored Clinical Resources for Promoting Children's Healthy Food Preferences
Brief Title: Toddler Tastes Study
Acronym: TTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Stephanie Anzman-Frasca, Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00008595; 1UM1TR005296 (NIH)
Record Dates: First submitted 2025-03-04; First posted 2025-03-14 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Dietary Behavior
Keywords: food preferences; toddlers; associative conditioning; modeling; food fussiness; vegetable acceptance; dietary intake
MeSH Terms: conditions — Food Preferences; Food Fussiness

STUDY DESIGN:
Masking Description: Masking is not possible in this study, as participants will know which intervention they are experiencing, as will the staff member conducting outcome assessments. Randomization will not occur until after baseline measurements are collected, and a staff member who will not have any other role in the study determined the randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Associative conditioning (Veggie and Dip tastings) (Experimental): Child is offered a vegetable to taste with a palatable dip, over 8 occasions. Tastings occur at home with the parent serving the vegetable and following standard scripting.
  Interventions: Behavioral: Associative conditioning
- Modeling (Parent and Me tastings) (Experimental): Child is offered a vegetable to taste while their parent/caregiver also tastes it and models enjoying it, over 8 occasions. Tastings occur at home with the parent serving and tasting the vegetable following standard scripting.
  Interventions: Behavioral: Modeling

INTERVENTIONS:
Behavioral: Associative conditioning — Child is offered a vegetable to taste with a palatable dip, over 8 occasions. Vegetable is served at home by parent/caregiver following standard script.
  Arms: Associative conditioning (Veggie and Dip tastings)
Behavioral: Modeling — Child is offered a vegetable to taste while their parent/caregiver also tastes it and models enjoying it, over 8 occasions. Vegetable is served at home with parent/caregiver following standard scripting.
  Arms: Modeling (Parent and Me tastings)

SUMMARY:
The goal of this study is to determine the feasibility and acceptability of two food preference learning approaches for toddlers that could serve as alternatives to mere repeated exposure to new or previously disliked foods. The target population is toddlers who score higher on food fussiness.

The study is a two-group randomized controlled trial. Families will be randomized to 1 of 2 study groups: associative conditioning, or the child tasting vegetables alongside a palatable dip, or modeling, in which the child and parent taste vegetables together. Both groups will attend two laboratory visits, one before and one after a 4-week exposure period, and will be asked to complete 8 vegetable tastings in accordance with their assigned condition across the 4 intervention weeks.

Key questions to be addressed are:

* summarizing the feasibility and acceptability of the intervention strategies
* assessing whether children's liking and intake of the target food increase from baseline to post-intervention

DETAILED DESCRIPTION:
Repeated exposure is a food preference learning strategy with a large evidence base, but there is a deficit in the literature regarding its effectiveness for children higher in food fussiness. The goal of this research is to identify strategies for young children who might need alternatives to repeated exposure to help them learn to accept vegetables. The approaches that will be evaluated are modeling and associative conditioning, and it is hypothesized that in both groups, children will show greater liking and intake of their target food post-intervention compared to baseline. Group differences in this potential increase, as well as feasibility and acceptance of the intervention strategies among the target population will be explored and summarized.

The study will be interventional. Families, stratified by child age and sex, will be randomized to 1 of 2 study groups: associative conditioning or modeling. Both groups will attend two laboratory visits, one baseline and one post-intervention assessment, and between these will complete 8 target vegetable taste exposures across 4 intervention weeks.

During screening, parents will be asked questions that will inform selection of their child's target vegetable (and dip if applicable). Using 3 vegetables from the literature, parents will report on whether they have served each of those vegetables, whether their child tasted it, and whether they would like their child to eat that vegetable. One of these vegetables will be chosen as the target vegetable to be tasted by the child during the study. The goal is to assign a vegetable that the child could use help learning to like/eat, that the parent would also like to serve at home. During screening, parents will also be asked to rate their child's liking of specific dips, which will inform which dip is provided to those that are assigned to the associative conditioning group (i.e. a dip they are likely to enjoy will like). Vegetables, and dips if applicable, will be provided.

After screening, a ~1 hour baseline laboratory visit will be scheduled. During the visit, written informed consent (parent) and verbal assent (child) will be completed. The child will be able to play with toys in the waiting room with the research staff and parent prior to the assent procedures to allow the child to acclimate to the environment and staff. Children will then be told that it is time to taste foods, and that they will come to a different room, with study staff and their parent, if they would like to do this activity. Vegetables will then be served to children (without any accompaniments/dip or modeling), and children's liking and intake will be measured via parent perceptions of liking and weighed plate waste, respectively. The child will be asked to try a bite of the vegetable. Then one-half cup of the study vegetable will be provided to the child, and they will be told they can eat as much or as little of the vegetable as they like. Parents will be asked to rate how much they think their child liked the vegetable, and the vegetable will be pre and post weighed to indicate consumption. At this visit, parents will also complete a survey that includes questions about demographics. At the end of the session, families will be randomized (i.e., associative conditioning or modeling groups) and provided with the intervention materials needed to complete the at-home exposures, including the target vegetable, instructions, and dips if applicable. Study staff will provide and explain the activity materials to families. Parents will be given opportunities to ask any questions, and staff will be trained to provide guidance and help problem solve implementation barriers as needed.

During the 4-week intervention period, parents will complete 2 exposures per week (8 total). During exposures, children in the associative conditioning group will be served a target vegetable with a liked dip. In the modeling group, a target vegetable will be served to both parent and child, with specific instructions provided to the parent on how to taste and react to the vegetable. Text reminders will be sent prior to each week to remind parents about the exposures. Parents will also complete brief, <5 minute online surveys at the end of each week. Surveys will assess whether the tastings were implemented as assigned, whether the child tasted/ate the vegetable, and parent perceptions of the child's liking of the vegetable.

Following the 4-week intervention period, families will attend a post-intervention assessment in the lab (~1 hr). Children's liking and intake of the target will be assessed as at baseline. The target vegetable will be served without dip or modeling, as at baseline, and parents will complete an audio-recorded, structured interview regarding their thoughts on the program they received during the study, strategies they use to feed their child, and views on potential clinical tools that could be used by pediatricians to communicate with families about increasing acceptance of healthy foods. Study staff will play with the child with toys in the waiting area while the parent completes the interview.

Approximately 40 parent-child dyads will be enrolled, with approximately half of the sample randomly assigned to the associative conditioning group and half to the modeling group, stratifying on child sex and age. Feasibility and acceptability will be summarized using descriptive statistics (survey data) and thematic analysis (interview data). Outcomes include the percentage of assigned tastings that were implemented as intended and whether this varies by group or individual or family characteristics. Parent feedback including barriers and facilitators to implementing programs will be summarized, as well as refinements that may improve the programs. Paired samples t-tests will test whether children's liking and intake of the target food increase from baseline to post-test (or an analogous non-parametric test if appropriate) overall; potential group differences in these changes will also be tested.

ELIGIBILITY:
Note: Age limits above reflect parents and children combined. Maximum age for children is 36 months as indicated below, and minimum age for parents/guardians is 18 years.

Inclusion Criteria:

* Child is 18-36 months old
* Parent/guardian is 18 years of age or older
* Parent/guardian participating is the primary caregiver of the child
* Child is not diagnosed with a physical or mental health condition (e.g., allergies to study foods, ARFID or autism diagnosis) that would impact safe or feasible participation
* Participants are English speakers
* Child is high on food fussiness, defined as a 2.5 or above on the food fussiness scale of the Child Eating Behavior Questionnaire for toddlers

Exclusion Criteria:

* The child is outside the age range of 18-36 months at enrollment, as verified by birth date
* Child is diagnosed with a physical or mental health condition that precludes safe or feasible participation
* The parent/guardian is less than 18 years old
* The parent/guardian participating is not the primary caregiver of the child
* Participants are not English speakers
* Child is low on food fussiness, defined as below a 2.5 on the food fussiness scale of the Child Eating Behavior Questionnaire for toddlers

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of the food preference learning approaches | Intervention (Weeks 1-4 after baseline assessment)
  Parents/guardians (here forward parents) will report on whether target food tastings were implemented as assigned. A percentage of assigned tastings that were implemented will be calculated (number of completed tastings divided by 8).
Acceptability of the food preference interventions | Intervention (Weeks 1-4 after baseline assessment)
  Themes from parent interviews will be summarized to inform how acceptable the study sample found each intervention.

SECONDARY OUTCOMES:
Change in vegetable liking | Baseline, post-intervention (Week 5)
  Changes in parent-reported child liking of the assigned study vegetable from baseline to post-intervention will be calculated. Liking is measured using a visual analog scale along which parents report how much they think the child enjoyed the served food on a scale of 1 to 9 where 1 is disliked extremely and 9 is liked extremely.
Change in vegetable intake | Baseline, post-intervention (Week 5)
  Changes in intake of the study vegetable will be calculated from baseline to post-intervention using weighed plate waste (weight of vegetable at post-intervention minus weight at baseline).

CONTACTS AND LOCATIONS:
Locations (1):
- Child Health and Behavior Lab at the University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be shared upon reasonable request after planned analyses are completed by the study team.